CLINICAL TRIAL: NCT06755775
Title: PET Imaging Targeting Granzyme B Predicts Immunotherapy Efficacy in Diffuse Large B-cell Lymphoma
Status: Recruiting | Type: Observational
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, LI BIAO, chief physician, Ruijin Hospital
Other Study IDs: RuijinH 2024-254
Record Dates: First submitted 2024-12-17; First posted 2025-01-01 (Actual); Last update posted 2025-01-01 (Actual); Status verified 2024-12

CONDITIONS: Diffuse Large B-Cell Lymphoma
Keywords: PET/CT; Granzyme B; immunotherapy
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lipodystrophy, Congenital Generalized

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- patients diagnosed with DLBCL who will receive immunotherapy (CAR-T, glofitamab, iR2)

SUMMARY:
This study aims to investigate the predictive value of PET imaging targeting granzyme B on the outcome of patients with diffuse large B lymphoma receiving immunotherapy.

DETAILED DESCRIPTION:
The investigators will number all participants, create a medical record file, and record their basic information (gender, age) as well as contact information and medical history information. All participants will undergo 68Ga-grazytracer PET at baseline and after one course of immunotherapy (CAR-T, Glofitamab or iR2 ).

ELIGIBILITY:
Inclusion Criteria:

1. Pathologic diagnosis of DLBCL
2. Patient's general condition is good and survival is expected to be greater than six months
3. Signed and dated informed consent form

Exclusion Criteria:

1. Combined with other malignant tumors
2. Patients with serious medical conditions who, in the opinion of the investigator, are not suitable for participation in this clinical study
3. Pregnant women and women at risk of pregnancy, breastfeeding women
4. poor compliant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chinese patient with pathologically confirmed diffuse large B-cell lymphoma
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-07-23 (Actual); Primary Completion 2029-07-23 (Estimated); Study Completion 2029-07-23 (Estimated)

PRIMARY OUTCOMES:
The value of PET imaging targeting granzyme B in predicting the efficacy of immunotherapy for diffuse large B-cell lymphoma | Baseline and 2 weeks after treatment
  The value of PET imaging targeting granzyme B in predicting the efficacy of immunotherapy for diffuse large B-cell lymphoma
Standardized uptake value (SUV) | Baseline and 2 weeks after treatment
  SUV of 68Ga-grazytracer uptake on PET/CT images for tumor lesions

SECONDARY OUTCOMES:
Progress free suivival | 3 years
  Progress free suivival
Overall survival | 3 years
  Overall survival

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital Affiliated to Shanghai Jiao Tong University Medical School, Shanghai, China

IPD SHARING:
Plan to Share IPD: No